CLINICAL TRIAL: NCT03691181
Title: Home COPD and Open Ventilation Evaluation (HOPE) Study
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landon Pediatric Foundation (Other)
Collaborators: Breathe Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study 210: H.O.P.E.
Record Dates: First submitted 2017-07-05; First posted 2018-10-01 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Outpatient ventilator support
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Open Ambulatory Ventilation (Experimental): monitoring with the use of the Life2000 Open Ventilation System for a period of six months with measures of nutrition, feeling of breathlessness, exercise tolerance, and quality of life.
  BODE Index B - BMI - BMI stands for body mass index, a calculation made by comparing height vs weight.
  O - Airway obstruction - Airway obstruction is measured by evaluating FEV1 - the amount of air that can be forcefully exhaled in 1 second after a deep breath.
  D - Dyspnea - Dyspnea refers to the degree of breathlessness someone experiences while living with COPD.
  E - Exercise tolerance - Exercise testing refers to how well some does on a 6-minute walk test.
  Modified Medical Research Council Dyspnea Scale
  Interventions: Device: Ventilation

INTERVENTIONS:
Device: Ventilation — monitoring with the use of the Life2000 Ventilation System for a period of six months
  Other Names: Ambulatory

SUMMARY:
Respiratory related diseases such as chronic obstructive pulmonary disease (COPD) and neuromuscular diseases remain a major public health issue affecting millions of people worldwide. More than 15 million people are estimated to be diagnosed with COPD in the US alone. In the US, the direct and indirect costs associated with COPD are estimated to be about $50 billion. Clinical studies have shown that by providing ventilation to reduce respiratory insufficiency symptoms such as dyspnea, patients may become more tolerant to exercise and be able to increase their participation in activities of daily living resulting in an overall positive impact in their quality of lives. The Life2000 Ventilation System, with the smallest tubing and comfortable interface solutions, is the only ventilator to simultaneously provide full ventilatory support and enable patients to ambulate.

The Life2000 Ventilation System is an FDA-cleared critical care ventilator (K141943/S003, June 2015) indicated for use for adult patients who require positive pressure ventilation delivered invasively or non-invasively. The device, classified by FDA as a continuous ventilator, can treat both acute and chronic respiratory failure and is suitable for use in home and institutional settings by qualified, trained personnel under the direction of a physician.

The Life2000 Compressor is intended to provide a 50-psi pressure source to the ventilator and is currently in the FDA premarket notification (510 k) clearance process, so its use is considered investigational.

DETAILED DESCRIPTION:
This will be a single-center, open-label, pilot study in 10 stable COPD subjects to assess the ventilatory efficacy of the Life2000 Ventilation System, as compared to a control group. Other important secondary endpoints as listed in this document will also be measured and reported. Prospective participants are all current participants in the ongoing CATCH program study. Subjects will be randomized to either continued monitoring alone or monitoring with the use of the Life2000 Ventilation System for a period of six months.

Initial BODE Index (BMI, airway Obstruction, Dyspnea, Exercise intolerance), CO2 (carbon dioxide) measurements, and questionnaires and surveys are captured prior to therapy initiation. Thereafter, subjects will be randomly assigned to the Life2000 Ventilation System or their routine plan of care, as determined previously by the CATCH program, and followed for a period of six months. Both end tidal CO2 readings and the Physical Activity Scale for the Elderly (PASE) results will be captured at pre-assigned intervals during the study. Monthly phone assessments will be conducted with the subjects to track progress. An additional BODE Index measurement will be taken at Day 90, the study mid-point. At the end of six months, all baseline procedures and questionnaires will be repeated and the subject will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:• Enrollment in the CATCH Study program

* Adults 40 years and older, as per inclusion criteria of the CATCH study
* Subjects with diagnosis of COPD (with and without chronic respiratory failure)
* Gold 3 & 4
* Ability and willingness to correctly execute and comply with study requirements

  o Ability and willingness to use the Life2000 Ventilation System a minimum of 6 hours/day (24 hr period).
* Requirement of supplemental oxygen to maintain an SpO2 > 88% at rest or during exercise
* Acceptable health status as assessed by medical history and/or physical exam
* Fluency in written and spoken English language
* Provision of written informed consent to participate in the study

Exclusion Criteria:• History of pneumothorax secondary to lung bullae

* Musculoskeletal or other non-pulmonary impairment that limits exercise tolerance
* Intolerance or unwillingness to utilize the Life2000 Ventilation System
* Women who are pregnant or nursing a child
* Presence of any condition or abnormality that in the opinion of the principal investigator may compromise the subject's safety or the quality of the study data

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
BODE Index change | 6 months
  Score can range from 0 to 10. Higher score is associated with increased survival.
  B - Body Mass Index Values 0 points for a BMI greater than 21 1 point for a BMI less than 21 O - Airway Obstruction Values 0 points for an FEV1 greater than 64%
  1 point for an FEV1 of 50-64% 2 points for an FEV1 of 36-49% 3 points for an FEV1 of less than 36% D - Dyspnea Values 0 points for a dyspnea index of 0-1
  1. point for a dyspnea index of 2
  2. points for a dyspnea index of 3
  3. points for a dyspnea index of 4-5 E - Exercise Tolerance Values
  0 point if able to walk over 349 meters
  1. point if able to walk 250-249 meters
  2. points if able to walk 150-249 meters
  3. points if able to walk 150 meters or less

SECONDARY OUTCOMES:
pre vs. on-ventilator days' change | 6 months
  Secondary endpoints will compare mean pre vs. on-ventilator days' differences in:
Borg Dyspnea Scale - | prior to start of therapy, upon therapy initiation, and again at Days 1, 30, 90, and 180.
  Borg scale a numerical scale for assessing dyspnea, from 0 representing no dyspnea to 10 as maximal dyspnea.
VENTILATOR USAGE | Monthly for six months
  Average daily ventilator usage (acquired during monthly phone questionnaire)
PASE | prior to therapy initiation (baseline) and again at Days 30, 90, and 180.
  Physical Activity Scale for the Elderly (PASE) - Physical Activity Scale for the Elderly (PASE) is a brief (5 minutes) and easily scored survey designed specifically to assess physical activity in epidemiological studies of persons age 65 years and older.The PASE score combines information on leisure, household and occupational activity. High Score is associated with good health.
HEALTH CARE COSTS | Six months prior to initiation and at 180 days
  Change in healthcare utilization and costs. Examples of healthcare utilization parameters would include emergency room visits and/or hospitalizations due to exacerbations and unscheduled office visits

CONTACTS AND LOCATIONS:
Locations (1):
- VCMC, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No